CLINICAL TRIAL: NCT05295004
Title: The Effect of Mindfulness Training Before Primary Total Joint Arthroplasty on Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Jason Jennings, Orthopedic Surgeon, Colorado Joint Replacement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1845025
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Sleep Disturbance; Arthropathy
MeSH Terms: conditions — Parasomnias; Joint Diseases

STUDY DESIGN:
Intervention Model Description: Randomize à Arm 1 (No Treatment), Arm 2 (Mindfulness Video @ Pre-Op), Arm 3 (Mindfulness Video @ Pre-Op, 1 Day Prior to surgery, 3 day's Post OP, 2 Weeks Post OP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Treatment (No Intervention): Patient will receive no mindfulness meditation training.
- Mindfulness at Pre-Op (Experimental): Patient will receive a one time training at their pre-operative appointment.
  Interventions: Behavioral: Mindfulness Meditation Training
- Multiple Mindfulness Meditation (Experimental): Mindfulness Video Training at Pre-Op, 1 Day Prior to surgery, 3 day's Post OP and 2 Weeks Post OP.
  Interventions: Behavioral: Mindfulness Meditation Training

INTERVENTIONS:
Behavioral: Mindfulness Meditation Training — Patient will watch a 10 minute video on how to use mindfulness meditation to help with sleep after a total joint replacement procedure.
  Arms: Mindfulness at Pre-Op; Multiple Mindfulness Meditation

SUMMARY:
The primary purpose of this study is the determine whether a 15 minute Mindfulness Meditation (MM) administered at the preoperative appointment prior to primary unilateral total joint arthroplasty (TJA) results in any improvement in Pittsburg Sleep Quality Index (PSQI) score, a validated metric for sleep quality, at 2, 6 or 12 weeks post-operatively.

DETAILED DESCRIPTION:
The primary purpose of this study is the determine whether a 15 minute Mindfulness Meditation (MM) administered at the preoperative appointment prior to primary unilateral total joint arthroplasty (TJA) results in any improvement in Pittsburg Sleep Quality Index (PSQI) score, a validated metric for sleep quality, at 2, 6 or 12 weeks post-operatively. We hypothesize that patients in the MM cohort will have lower PSQI scores, indicating higher sleep quality, at both post-operative time points. Secondary aims include characterizing differences between cohorts in Visual Analog Scale (VAS) for pain, Epworth Sleepiness Scale (ESS) scores, Patient Reported Outcome Measurement Information System - Sleep Disturbance - Short Form, and Knee Injury and Osteoarthritis Outcome Scores (KOOS) at 2, 6 and 12 weeks following TJA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total joint arthroplasty at Colorado Joint Replacement
* Between the ages of 18 and 90 years old will be included in the study.

Exclusion Criteria:

* Simultaneous total joint arthroplasty
* Uni-compartmental knee arthroplasty
* Revision surgery for infection, fracture or other indication.
* History of Drug or Alcohol Abuse
* Patients who are unable to present at a standard pre-operative appointment within 4 weeks prior to scheduled surgery will also be excluded, as the MM intervention would not be possible to administer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index score | Change from Pre-Op to 2, 6 and 12 weeks post op.
  Improvement in Pittsburg Sleep Quality Index (PSQI) score, Scale is 0 to 21, higher score is worse outcome.

SECONDARY OUTCOMES:
Visual Analog Score | Change from Pre-Op to 2, 6 and 12 weeks post op.
  Improvement in Visual Analog Score (VAS), Scale is 1 to 10, higher score is worse outcome
Epworth Sleepiness Scale | Change from Pre-Op to 2, 6 and 12 weeks post op.
  Improvement in Epworth Sleepiness Scale (ESS), Scale is 0 to 24, higher score is worse outcome
Knee Injury and Osteoarthritis Outcome Scores JR | Change from Pre-Op to 2, 6 and 12 weeks post op.
  Improvement in Knee Injury and Osteoarthritis Outcome Scores JR (KOOS JR), Scale is 1 to 100, lower score is worse outcome
Knee Society Score (KSS) | Change from Pre-Op to 6 Weeks post op.
  Improvement in Knee Society Score (KSS), Scale is 0 to 100, lower score is worse outcome
Patient Reported Outcome Measurement Information System - Sleep Disturbance (PROMIS-SD) | Change from Pre-Op to 2, 6 and 12 weeks post op.
  Improvement in Patient Reported Outcome Measurement Information System - Sleep Disturbance (PROMIS-SD), Scale is 8 to 40, higher score is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Jennings, MD, DPT, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

REFERENCES:
- [Result] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Result] Chen AF, Orozco FR, Austin LS, Post ZD, Deirmengian CA, Ong AC. Prospective Evaluation of Sleep Disturbances After Total Knee Arthroplasty. J Arthroplasty. 2016 Jan;31(1):330-2. doi: 10.1016/j.arth.2015.07.044. Epub 2015 Aug 30. PMID 26455403
- [Result] Er MS, Altinel EC, Altinel L, Erten RA, Eroglu M. An assessment of sleep quality in patients undergoing total knee arthroplasty before and after surgery. Acta Orthop Traumatol Turc. 2014;48(1):50-4. doi: 10.3944/AOTT.2014.3163. PMID 24643100
- [Result] Chhangani BS, Roehrs TA, Harris EJ, Hyde M, Drake C, Hudgel DW, Roth T. Pain sensitivity in sleepy pain-free normals. Sleep. 2009 Aug;32(8):1011-7. PMID 19725252
- [Result] Manrique J, Gomez MM, Parvizi J. Stiffness after total knee arthroplasty. J Knee Surg. 2015 Apr;28(2):119-26. doi: 10.1055/s-0034-1396079. Epub 2014 Dec 16. PMID 25513992
- [Result] Dowsey M, Castle D, Knowles S, Monshat K, Salzberg M, Nelson E, Dunin A, Dunin J, Spelman T, Choong P. The effect of mindfulness training prior to total joint arthroplasty on post-operative pain and physical function: A randomised controlled trial. Complement Ther Med. 2019 Oct;46:195-201. doi: 10.1016/j.ctim.2019.08.010. Epub 2019 Aug 12. PMID 31519279
- [Result] Hanley AW, Gililland J, Erickson J, Pelt C, Peters C, Rojas J, Garland EL. Brief preoperative mind-body therapies for total joint arthroplasty patients: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1749-1757. doi: 10.1097/j.pain.0000000000002195. PMID 33449510
- [Result] Kiran U, Ladha S, Makhija N, Kapoor PM, Choudhury M, Das S, Gharde P, Malik V, Airan B. The role of Rajyoga meditation for modulation of anxiety and serum cortisol in patients undergoing coronary artery bypass surgery: A prospective randomized control study. Ann Card Anaesth. 2017 Apr-Jun;20(2):158-162. doi: 10.4103/aca.ACA_32_17. PMID 28393774
- [Result] Packiasabapathy S, Susheela AT, Mueller A, Patxot M, Gasangwa DV, O'Gara B, Shaefi S, Marcantonio ER, Yeh GY, Subramaniam B. Guided meditation as an adjunct to enhance postoperative recovery after cardiac surgery: study protocol for a prospective randomized controlled feasibility trial. Trials. 2019 Jan 11;20(1):39. doi: 10.1186/s13063-018-3103-8. PMID 30635064
- [Result] Chavez JL, Porucznik CA, Gren LH, Guan J, Joyce E, Brodke DS, Dailey AT, Mahan MA, Hood RS, Lawrence BD, Spiker WR, Spina NT, Bisson EF. The Impact of Preoperative Mindfulness-Based Stress Reduction on Postoperative Outcomes in Lumbar Spine Degenerative Disease: 3-Month and 12-Month Results of a Pilot Study. World Neurosurg. 2020 Jul;139:e230-e236. doi: 10.1016/j.wneu.2020.03.186. Epub 2020 Apr 9. PMID 32278820
- [Result] Ong JC, Manber R, Segal Z, Xia Y, Shapiro S, Wyatt JK. A randomized controlled trial of mindfulness meditation for chronic insomnia. Sleep. 2014 Sep 1;37(9):1553-63. doi: 10.5665/sleep.4010. PMID 25142566
- [Result] Rusch HL, Rosario M, Levison LM, Olivera A, Livingston WS, Wu T, Gill JM. The effect of mindfulness meditation on sleep quality: a systematic review and meta-analysis of randomized controlled trials. Ann N Y Acad Sci. 2019 Jun;1445(1):5-16. doi: 10.1111/nyas.13996. Epub 2018 Dec 21. PMID 30575050
- [Result] Shakya H, Wang D, Zhou K, Luo ZY, Dahal S, Zhou ZK. Prospective randomized controlled study on improving sleep quality and impact of zolpidem after total hip arthroplasty. J Orthop Surg Res. 2019 Sep 3;14(1):289. doi: 10.1186/s13018-019-1327-2. PMID 31481074